CLINICAL TRIAL: NCT03750331
Title: Impact of the Use of Remote Monitoring in the Follow-up of the Renal Transplant Patient.
Acronym: APT'x
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1708232; 2018-A00677-48 (Other: ID-RCB)
Record Dates: First submitted 2018-11-08; First posted 2018-11-23 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Renal Transplantation
Keywords: telemedicine

STUDY DESIGN:
Intervention Model Description: Non-inferiority Randomized Controlled Trial comparing Non-inferiority Randomized Controlled Trial comparing (i) a group of renal transplant outpatients consulting their Transplant Centre following a traditional schedule (every other week up to 6 months post-transplant, once a month up to year 1, every three months up to year 2 and every 6 months thereafter) to (ii) a group of patients assisted by Ap'TELACARE and consulting their Transplant Centre following a less stringent schedule of consultations (every month up to 6 months, every other month up to year 1, every six months up to year 2 and once a year thereafter).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional patient follow-up (Active Comparator): a group of renal transplant outpatients consulting their Transplant Centre following a traditional schedule (every other week up to 6 months post-transplant, once a month up to year 1, every three months up to year 2 and every 6 months thereafter)
  Interventions: Other: traditional schedule
- medically-tailored follow-up with Ap'Telecare (Experimental): a group of patients assisted by Ap'Telecare and consulting their Transplant Centre following a less stringent schedule of consultations (every month up to 6 months, every other month up to year 1, every six months up to year 2 and once a year thereafter).
  Interventions: Other: Ap'Telecare

INTERVENTIONS:
Other: Ap'Telecare — an internet application on a computer, tablet or smartphone
  Arms: medically-tailored follow-up with Ap'Telecare
Other: traditional schedule — a group of renal transplant outpatients consulting their Transplant Centre following a traditional schedule
  Arms: traditional patient follow-up

SUMMARY:
Transplant Centers are facing new organisational challenges with regards to the growing number of patients they have to follow-up. We have developed and assessed the feasibility of using a novel web application permitting a medically-tailored follow-up of stable renal transplanted outpatients: Ap'TELECARE. This novel approach is likely to facilitate the organization of patients' follow-up at the Transplant Centre level as well as to provide secondary individual benefits in terms of therapeutic education, adherence to treatment and eventually to improve long term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted for at least 3 months
* Stable renal graft function

Exclusion Criteria:

* No home internet access
* Major disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 738 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patients experiencing at least one episode of graft dysfunction | 2 years
  graft dysfunction defined by a drop of at least 20% of their usual estimated Glomerular Filtration Rate (eGFR) value)

SECONDARY OUTCOMES:
Failure of immunosuppressive treatment | 2 years
  Detection of donor-specific anti-HLA (Human Leukocyte Antigen) antibodies by LUMINEX technic
number of patients who needed to return to dialysis | 2 years
number of patients with acute or chronic transplant rejection | 2 years
Post-transplant complication | 2 years
Death | 2 years
Quality of life assessed | 2 years
  EuroQol group - 5 Dimensions ( EQ-5D) scale
Level of anxiety and depression | 2 years
  Hospital Anxiety and Depression (HAD) scale
Incremental cost-effectiveness evaluation criteria | 2 years
  Cost per QALY earned (QALYs estimated from the EuroQol group - 5 Dimensions ( EQ-5D) quality of life scale).
Evaluation criteria for the Budget Impact Analysis | 2 years
  Average cost saved per 100 patients treated in the "Ap'Telecare group" compared to the "traditional follow-up".

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Mariat, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Clermont-Ferrand, CHU Site Gabriel-Montpied, Clermont-Ferrand
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No